CLINICAL TRIAL: NCT01603420
Title: Phase 2/3 Study of Dose-escalated External Beam Radiation Therapy With or Without Chemotherapy for High Risk Adenocarcinoma of the Prostate
Brief Title: External Beam Radiation With or Without Chemotherapy to Treat High Risk Prostate Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: enrollment goals not met
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GU004-11
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; radiation; proton; chemotherapy; high risk
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Gonadotropin-Releasing Hormone; Goserelin; Leuprolide; luprolide acetate gel depot; Docetaxel; Radiotherapy, Intensity-Modulated; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation + 24mo luteinizing hormone-releasing hormone (LHRH) (Active Comparator): Conformal RT 79.2 Gy(RBE) total dose + 24 months LHRH agonist (androgen suppression).
  Interventions: Drug: Luteinizing hormone-releasing hormone (LHRH); Other: Conformal Radiation Therapy (RT)
- Radiation + Chemo + 6mo luteinizing hormone-releasing hormone (Experimental): Conformal RT 79.2 Gy(RBE) total dose + Chemotherapy: Docetaxel 20mg/m2 x every 7 days x 8 weeks followed by 6 months LHRH (androgen suppression).
  Interventions: Drug: Luteinizing hormone-releasing hormone (LHRH); Drug: Docetaxel; Other: Conformal Radiation Therapy (RT)

INTERVENTIONS:
Drug: Luteinizing hormone-releasing hormone (LHRH) — Androgen suppression therapy using luteinizing hormone-releasing hormone (LHRH) agonists such as leuprolide, goserelin, buserelin, triptorelin.
  Other Names: -Androgen Suppression; -Androgen Deprivation; -Zoladex; -Lupron; -Eligard; -Viadur
Drug: Docetaxel — Docetaxel 20mg/m2 IV every 7 days x 8 weeks.
  Other Names: -taxotere; -docetaxel
  Arms: Radiation + Chemo + 6mo luteinizing hormone-releasing hormone
Other: Conformal Radiation Therapy (RT) — 1.8 Gy(RBE) (or Gy for IMRT) per fraction,five fractions per week for a total dose of 79.2 Gy (RBE) (or Gy).
  Other Names: Intensity-modulated Radiation Therapy (IMRT); Proton Therapy; Particle Therapy

SUMMARY:
The purpose of this study is to compare the effects on prostate cancer using radiation therapy with or without chemotherapy.

DETAILED DESCRIPTION:
The recommended treatment for a high risk prostate cancer consists of a combination of radiation therapy and androgen suppression for 2-3 years. Recent studies have shown a survival advantage for chemotherapy for prostate cancer. Chemotherapy has already been successfully integrated in the treatment of other cancer types and is our belief that chemotherapy will prove to be beneficial for patients with high risk prostate cancer. However, a clinical study is necessary to compare the results good or bad of chemotherapy with radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma (within 365 days of randomization.
* High-risk for recurrence as determined by evidence of at least one of the following: Gleason score 8-10, PSA > 20, T state T3.
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material: Gleason score must be in the range 2-10. > 6 cores are strongly recommended.
* Clinical stages T1a- T3 N0 M0 as staged by the treating investigator. (AJCC Criteria 7th Ed.-appendix III).
* PSA values < = 50 ng/ml within 90 days prior to randomization. Must be completed prior to biopsy or at least 21 days after prostate biopsy.
* Absolute Neutrophil Count (ANC) > = 1,800 cells/mm³ within 90 days prior to randomization.
* Platelets > = 100,000 cells/mm³ within 90 days prior to randomization.
* Hemoglobin > 10 g/dl within 90 days prior to randomization.
* ALT, AST, and total bilirubin within 1.5 X institutional upper normal limits within 90 days prior to randomization.
* ECOG status 0-1 (appendix II) documented within 90 days of randomization.
* Patient must sign study specific informed consent prior to randomization. Note: consent for legally authorized representative is not permitted.
* Completed all requirements listed in section 4.0 within the specified time frames.
* Able to start treatment within 56 days of randomization.
* At least 18 years old and less than or equal to 75 years of age.
* Men of child-producing potential must be willing to consent to use effective contraception while on treatment and for at least 3 months afterwards.
* Medical oncology consultation prior to randomization and medically approved for chemotherapy treatment per protocol.

Exclusion Criteria:

* Evidence of distant metastasis.
* Pelvic lymph nodes > 1.5 cm in greatest dimension unless the enlarged lymph node is biopsied and negative.
* Prior prostate cancer surgery including but not limited to prostatectomy, hyperthermia and cryosurgery.
* Prior pelvic radiation for their prostate cancer.
* Prior androgen deprivation.
* Severe, active co-morbidity, defined as follows:
* Active rectal diverticulitis, Crohn's disease affecting the rectum or ulcerative colitis. (Non-active diverticulitis and Crohn's disease not affecting the rectum are allowed).
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
* Myocardial infarction within the last 6 months.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of randomization.
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
* Prior allergic reaction to the drugs involved in this protocol.
* Existing peripheral neuropathy > = grade 2.
* Prior systemic chemotherapy for prostate cancer.
* History of proximal urethral stricture requiring dilatation.
* Major medical, addictive or psychiatric illness which in the investigator's opinion, will prevent the consent process, completion of the treatment and/or interfere with follow-up.
* Evidence of any other cancer within the past 5 years and < 50% probability of a 5 year survival. (Prior or concurrent diagnosis of basal cell or non-invasive squamous cell cancer of the skin is allowed.)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Vargas, MD, Study Chair — Proton Collaborative Group
Locations (3):
- United States (3):
  - CDH Proton Center, Warrenville, Illinois
  - Procure Proton Therapy Center, Oklahoma City, Oklahoma
  - Hampton University Proton Therapy Institute, Hampton, Virginia

REFERENCES:
- [Derived] Guttilla A, Bortolus R, Giannarini G, Ghadjar P, Zattoni F, Gnech M, Palumbo V, Valent F, Garbeglio A, Zattoni F. Multimodal treatment for high-risk prostate cancer with high-dose intensity-modulated radiation therapy preceded or not by radical prostatectomy, concurrent intensified-dose docetaxel and long-term androgen deprivation therapy: results of a prospective phase II trial. Radiat Oncol. 2014 Jan 14;9:24. doi: 10.1186/1748-717X-9-24. PMID 24423462

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation + 24mo LHRH: Conformal RT 79.2 Gy(RBE) total dose + 24 months LHRH agonist (androgen suppression).
  LHRH: Androgen suppression therapy using LHRH agonists such as leuprolide, goserelin, buserelin, triptorelin.
  Conformal RT: 1.8 Gy(RBE) (or Gy for IMRT) per fraction,five fractions per week for a total dose of 79.2 Gy (RBE) (or Gy).
- Radiation + Chemo + 6mo LHRH: Conformal RT 79.2 Gy(RBE) total dose + Chemotherapy: Docetaxel 20mg/m2 x every 7 days x 8 weeks followed by 6 months LHRH (androgen suppression).
  Docetaxel: Docetaxel 20mg/m2 IV every 7 days x 8 weeks.
  Conformal RT: 1.8 Gy(RBE) (or Gy for IMRT) per fraction,five fractions per week for a total dose of 79.2 Gy (RBE) (or Gy).
Period: Overall Study
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 53 [53 to 53] | 72 [72 to 72] | 62.5 [53 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 2 - Assessment of Number of Freedom From Failure Events in the Chemotherapy Arm
Description: Measurement of Freedom from Failure i.e. the first occurence of clinical failure (local recurrence, regional recurrence, or distant metastasis), biochemical failure by the Phoenix definition (Prostate Specific Antigen [PSA] > = 2 ng/ml over the nadir PSA discounting bounces per the investigators discretion), or the start of salvage therapy including androgen deprivation.
  This study was terminated prior to the time frame of 2 years being reached. Therefore, this outcome was assessed at time of study closure (22 months).
Time Frame: No failures were reported at the time of study termination (22 months). This outcome was originally written to assess failure at 2 years. However, that end point was not reached.
Population: No failures were reported at the time of study termination (22 months). This outcome was originally written to assess failure at 2 years. However, that end point was not reached.
Measure: Number; unit: failure events
Arm/Group | Radiation + 24mo Luteinizing Hormone-releasing Hormone (LHRH) | Radiation + Chemo + 6mo Luteinizing Hormone-releasing Hormone
Number analyzed (Participants) | 1 | 1
failure events | 0 | 0

2. Primary Outcome: Phase 2 - Assessment of Number of Freedom From Failure Event Comparing Chemotherapy Arm to Standard Treatment Arm
Description: This endpoint will be examined if decision is made to not move forward with phase 3 study.
  This study was terminated prior to a decision being made about moving on to a phase 3 study. Therefore, this outcome was not assessed.
Time Frame: at 5 years
Arm/Group | Radiation + 24mo Luteinizing Hormone-releasing Hormone (LHRH) | Radiation + Chemo + 6mo Luteinizing Hormone-releasing Hormone
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Phase 2 - Cumulative Number of Incidences of Grade 3 or Higher Adverse Events.
Description: Assessment will be performed using CTCAE v4 criteria.
  This study was terminated prior to the time frame of 2 years being reached. Therefore, this outcome was assessed at time of study closure (22 months).
Time Frame: 2 years
Population: This study was terminated prior to the time frame of 2 years being reached. Therefore, this outcome was assessed at time of study closure (22 months).
Measure: Number; unit: events
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Number analyzed (Participants) | 1 | 1
events | 0 | 0

4. Primary Outcome: Phase 3 - Assessment of the Number of Freedom From Failure (FFF) Events Comparing the Chemotherapy Arm to the Standard Treatment Arm.
Description: The events for FFF will be the first occurence of clinical failure (local recurrence, regional recurrence, or distant metastasis), biochemical failure by the Phoenix definition (PSA > = ng/ml over the nadir PSA discounting bounces per the investigators discretion), or the start of salvage androgen deprivation.
  This study was terminated prior to a decision being made about moving on to a phase 3 study. Therefore, this outcome was not assessed.
Time Frame: at 5 years
Population: This study was terminated prior to a decision being made about moving on to a phase 3 study. Therefore, this outcome was not assessed.
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Assessment of Number of Grade 2 or Higher Genitourinary (GU) and Gastrointestinal (GI) Adverse Events
Description: Assessment will be performed using CTCAE v 4 criteria.
Time Frame: at 6 months
Measure: Number; unit: incidences
Arm/Group | Radiation + 24mo Luteinizing Hormone-releasing Hormone (LHRH) | Radiation + Chemo + 6mo Luteinizing Hormone-releasing Hormone
Number analyzed (Participants) | 1 | 1
incidences | 0 | 1

6. Secondary Outcome: Assessment of Number of GI and GU Adverse Events
Description: Descriptive measurements of frequency will be compiled.
  This study was terminated prior to the time frame of 3 years being reached. Therefore, this outcome was not assessed. Data were collected on toxicities up until study closure at 22 months. However, this timepoint was not indicated as a secondary objective in the protocol. Therefore, data was not analyzed at time of study closure.
Time Frame: at 3 years
Arm/Group | Radiation + 24mo Luteinizing Hormone-releasing Hormone (LHRH) | Radiation + Chemo + 6mo Luteinizing Hormone-releasing Hormone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Assessment of Total Number of Local/Distant Failures
Description: The total number of local/distant failures will be assessed.
Time Frame: at time of study closure (22 months)
Measure: Number; unit: participants
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

8. Secondary Outcome: Assessment of Impotence by Summation of Relative Scores for Sexual Function From the EPIC Quality of Life Instrument.
Description: unable to assess due to lack of data
Time Frame: Up to 10 years
Population: unable to assess due to study termination
Arm/Group | Radiation + 24mo Luteinizing Hormone-releasing Hormone (LHRH) | Radiation + Chemo + 6mo Luteinizing Hormone-releasing Hormone
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Assessment of Total Number of Salvage Androgen Deprivation Use With Comparison of Arms.
Description: The total number of subjects with salvage androgen deprivation use will be assessed.
Time Frame: At study closure (22 months)
Measure: Number; unit: participants
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

10. Secondary Outcome: Assessment of Total Number of Survival Events With Comparison of Group Arms
Description: The number of deaths in both arms will be assessed.
Time Frame: at study closure (22 months)
Measure: Number; unit: participants
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

11. Secondary Outcome: Assessment of Total Number of Biochemical Failure Events
Description: The number of biochemical failure events will be assessed on both arms.
Time Frame: at study closure (22 months)
Measure: Number; unit: participants
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

12. Secondary Outcome: Assessment of Quality of Life - Summation of Relative Scores From the EPIC Instrument.
Description: unable to assess due to lack of data
Time Frame: Up to 10 years
Population: unable to assess due to study termination
Arm/Group | Radiation + 24mo Luteinizing Hormone-releasing Hormone (LHRH) | Radiation + Chemo + 6mo Luteinizing Hormone-releasing Hormone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Radiation + 24mo LHRH | Radiation + Chemo + 6mo LHRH
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation + 24mo LHRH (N=1) | Radiation + Chemo + 6mo LHRH (N=1)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
agitation (Psychiatric disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
hot flashes (Vascular disorders) | 1 (1) | 0 (0)
dermatitis radiation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No